CLINICAL TRIAL: NCT02384317
Title: An Open-Label Phase 2 Study to Evaluate the Safety and Efficacy of CCX168 in Subjects With Immunoglobulin A Nephropathy on Stable RAAS Blockade
Brief Title: Open-Label Study to Evaluate Safety and Efficacy of CCX168 in Subjects With IGA Nephropathy on Stable RAAS Blockade
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL005_168; 2014-003402-33 (EudraCT Number)
Record Dates: First submitted 2015-02-11; First posted 2015-03-10 (Estimated); Results first posted 2023-08-01 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Immunoglobulin A Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — avacopan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CCX168 (Avacopan) (Experimental): CCX168 (Avacopan) plus stable dose of RAAS blocker
  Interventions: Drug: CCX168

INTERVENTIONS:
Drug: CCX168 — CCX168 30 mg, twice daily (b.i.d.) orally for 84 days (12 weeks). The CCX168 dose was taken in the morning, optimally within one hour after breakfast, and in the evening, optimally within one hour after dinner.

SUMMARY:
The primary safety objective of this study is to evaluate the safety and tolerability of CCX168 in subjects with IgAN on background supportive therapy with a maximally tolerated dose of RAAS blockade. The primary efficacy objective is to evaluate the efficacy of CCX168 based on an improvement in proteinuria.

DETAILED DESCRIPTION:
Study acquired by Amgen and all disclosures were done by previous sponsor ChemoCentryx.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of Immunoglobulin A nephropathy
* estimated glomerular filtration rate >60 mL/min/1.73 m2
* Proteinuria (first morning urinary protein:creatinine ratio >1g/g creatinine)

Key Exclusion Criteria:

* Severe renal disease
* Pregnant or nursing
* Proteinuria >8g/g creatinine or >8g/day
* Systemic manifestations of Henoch-Schonlein purpura within 2 years prior
* Patients with Immunoglobulin A nephropathy deemed secondary to underlying disease
* Biopsy reported severe crescentic Immunoglobulin A nephropathy
* History of treatment with glucocorticoids, cyclophosphamide, azathioprine, mycophenolate mofetil, or any biologic immunomodulatory agent with 24 weeks prior
* History of clinically significant cardiac conditions
* History of cancer within 5 years prior
* Any infection requiring antibiotic treatment that has not cleared prior to study start

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-03-27 (Actual); Primary Completion 2015-09-13 (Actual); Study Completion 2018-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (6):
- United States (5):
  - Palo Alto, California
  - San Francisco, California
  - Reno, Nevada
  - Chapel Hill, North Carolina
  - Columbus, Ohio
- Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Screening took place for 14 days. Screening was following by a combined renin-angiotensin-aldosterone system (RAAS) titration (up to 4 weeks) plus run-in period (8 weeks) with an additional up to 7-day eligibility confirmation.
Groups:
- CCX168: Modified Intent-to-Treatment (mITT) Population included all subjects who received at least one dose of study drug and who had at least one post baseline urinary PCR assessment.
Period: Overall Study
Arm/Group | CCX168
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Safety Population included of all subjects who received at least one dose of study drug.
Arm/Group | Overall Study
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.1 (13.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4
  Sweden | 3
BMI [Mean (Standard Deviation); unit: kg/m²] — BMI = Body Mass Index
  kg/m² | 30.05 (8.29)
Mean time since diagnosis of IgAN [Mean (Full Range); unit: month] — IgAN = IgA Nephropathy
  month | 17.3 [1 to 42]
PCR [Mean (Full Range); unit: mg/g] — Urinary PCR = protein:creatinine ratio
  mg/g | 1906.84 [1181.06 to 3392.25]
ACR [Mean (Full Range); unit: mg/g] — Urinary ACR = Albumin to Creatinine Ratio
  mg/g | 1528.42 [921.76 to 2898.18]
eGFR [Mean (Full Range); unit: mL/min/1.73m²] — eGFR = estimated Glomerular Filtration Rate
  mL/min/1.73m² | 65.89 [48.91 to 93.91]
MCP-1 to Creatinine ratio [Mean (Full Range); unit: pg/mg crea] — MCP-1 = Monocyte Chemoattractant Protein-1
  pg/mg crea | 577.44 [224.79 to 974.70]

OUTCOME MEASURES:

1. Primary Outcome: Change in Slope of First Morning Urinary PCR From the 8-week RAAS Blocker run-in Period to the 12-week CCX168 Treatment Period
Description: The mean change in the slope of the urinary protein:creatinine ratio (UPCR, in mg/g/week) between the 8-week run-in period and the 12-week treatment period
Time Frame: Week -8 to -1 (Run-in period) and Week 1 to 12 (treatment period)
Measure: Mean (95% Confidence Interval); unit: mg/g/week
Groups:
- 8-week Run-in Period: 8-week RAAS run-in period
- 12-week Treatment Period: 12-week CCX168 treatment period
Arm/Group | CCX168 | 8-week Run-in Period | 12-week Treatment Period
Number analyzed (Participants) | 7 | 7 | 7
mg/g/week | -2.4 [-133.6 to 128.7] | 15.3 [-87.3 to 117.9] | -23.9 [-195.0 to 147.2]
Statistical Analysis 1: Comparison: 8-week Run-in Period vs 12-week Treatment Period; Test type: Superiority; p = 0.965, Random coefficients regression; Slope = -2.4, 95% CI 2-sided [-133.6 to 128.7], Standard Deviation 141.77

2. Primary Outcome: Number of Participants With AE's
Description: Acronyms use: Adverse Events (AE's) Serious Adverse Events (SAE's)
Time Frame: Day 0 - Day 169 (throughout the trial)
Measure: Count of Participants; unit: Participants
Groups:
- Safety Population: Safety Population included of all subjects who received at least one dose of study drug.
Arm/Group | Safety Population
Number analyzed (Participants) | 7
Participants
  Subjects who had any AE | 7
  Subjects who had an SAE | 1
  Subjects who had an AE possibly related | 5

3. Secondary Outcome: Proportion of Subjects Achieving Renal Response From Baseline to Day 85
Description: Renal Response defined as an improvement in proteinuria based on a decrease from baseline to Day 85 in proteinuria to a level <300 mg/g creatinine and maintaining eGFR within 15% of baseline.
Time Frame: Baseline and Day 85
Measure: Number; unit: proportion of participants
Arm/Group | CCX168
Number analyzed (Participants) | 7
proportion of participants
  Patients with a renal response by Day 85 | 0
  Patients with no renal response by Day 85 | 1

4. Secondary Outcome: Proportion of Subjects Achieving a Partial Renal Response From Baseline to Day 85
Description: A partial renal response, defined as an improvement in proteinuria based on a decrease from baseline to Day 85 in proteinuria to a level <1 g/g creatinine and maintaining eGFR within 15% of baseline.
Time Frame: Baseline and Day 85
Measure: Number; unit: proportion of participants
Arm/Group | CCX168
Number analyzed (Participants) | 7
proportion of participants
  Patients with a partial renal response at day 85 | 0.29
  Patients with no partial renal response at day 85 | 0.71

5. Secondary Outcome: Change From Baseline to Day 85 in Vital Signs
Time Frame: Baseline to day 85
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Safety Population
Number analyzed (Participants) | 7
beats per minute | 1.3 (8.56)

6. Primary Outcome: Severity of Adverse Events (AE's)
Description: Acronyms use: Adverse Events (AE's) Serious Adverse Events (SAE's)
Time Frame: Day 0 - Day 169 (throughout the trial)
Measure: Number; unit: Number of AEs
Arm/Group | Safety Population
Number analyzed (Participants) | 7
Number of AEs
  AE leading to interruption of treatment | 1
  AE leading to permanent discontinuation of study | 0
  Withdrawals due to AE | 0
  Deaths | 0
  AE of grade 3 ≥ | 1
  Related AE grade 3≥ | 0

7. Secondary Outcome: Change in Systolic Blood Pressure From Baseline to Day 85
Time Frame: Baseline to day 85
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Safety Population
Number analyzed (Participants) | 7
mmHg | -1.4 (12.11)

8. Secondary Outcome: Change in Diastolic Blood Pressure From Baseline to Day 85
Time Frame: Baseline to day 85
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Safety Population
Number analyzed (Participants) | 7
mmHg | 2.1 (8.45)

9. Secondary Outcome: Change in Temperature From Baseline to Day 85
Time Frame: Baseline to day 85
Measure: Mean (Standard Deviation); unit: C
Arm/Group | Safety Population
Number analyzed (Participants) | 7
C | 0.2 (0.68)

10. Secondary Outcome: Change in Weight From Baseline to Day 85
Time Frame: Baseline to day 85
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Safety Population
Number analyzed (Participants) | 7
kg | -0.6 (2.39)

ADVERSE EVENTS:
Time Frame: From Baseline up to 169 days
Groups:
- Safety Population: Safety population included all subjects who received any CCX168
Arm/Group | Safety Population
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 1/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Population (N=7)
Angina unstable (Cardiac disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population (N=7)
Headache (Nervous system disorders) | 3 (3)
Nasopharyngitis (Infections and infestations) | 3 (3)
Peripheral swelling (General disorders) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 2 (3)
Blood creatine phosphokinase increased (Investigations) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 2 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (4)
Nausea (Gastrointestinal disorders) | 2 (4)
Urinary tract infection (Infections and infestations) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Eosinophil count increased (Investigations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 1 (1)
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Localized oedema (General disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Parotitis (Infections and infestations) | 1 (1)
Polyuria (Renal and urinary disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Rhinovirus infection (Infections and infestations) | 1 (1)
Skin swelling (Skin and subcutaneous tissue disorders) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2015-07-17): https://cdn.clinicaltrials.gov/large-docs/17/NCT02384317/Prot_000.pdf
  • Statistical Analysis Plan (2016-10-03): https://cdn.clinicaltrials.gov/large-docs/17/NCT02384317/SAP_001.pdf